CLINICAL TRIAL: NCT05995600
Title: Comparison of Clopidogrel-based Antiplatelet Therapy Versus Warfarin As Secondary Prevention Strategy for AntiPhospholipid Syndrome-related STROKE (APS-STROKE)
Brief Title: Comparison of Clopidogrel-based Antiplatelet Therapy Versus Warfarin As Secondary Prevention Strategy for AntiPhospholipid Syndrome-related STROKE
Acronym: APS-STROKE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seung-Hoon Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2304-096-1425
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Antiphospholipid Syndrome; Ischemic Stroke; Transient Ischemic Attack; Cerebrovascular Disease; Cardiovascular Diseases; Major Bleed
Keywords: Antiphospholipid syndrome; Ischemic stroke; Secondary prevention; Thrombosis
MeSH Terms: conditions — Antiphospholipid Syndrome; Ischemic Stroke; Ischemic Attack, Transient; Cerebrovascular Disorders; Cardiovascular Diseases; Thrombosis | interventions — Platelet Aggregation Inhibitors; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective, Randomized, Open-label, Blinded Endpoint (PROBE) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clopidogrel-based antiplatelet therapy group (Experimental): Clopidogrel 75 mg daily
  Patients assigned to this group will be permitted to use additional antiplatelet drugs other than clopidogrel at the investigator's discretion.
  Interventions: Drug: Antiplatelet Drug
- Warfarin group (Active Comparator): Warfarin (target prothrombin time-international normalized ratio 2.0-3.0)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Antiplatelet Drug — Clopidogrel ± other antiplatelet drug
  Arms: Clopidogrel-based antiplatelet therapy group
Drug: Warfarin — Warfarin (target prothrombin time-international normalized ratio 2.0-3.0)
  Arms: Warfarin group

SUMMARY:
Antiphospholipid syndrome (APS) has a close association with ischemic stroke; however, the optimal treatment strategy for APS-related stroke has yet to be established. The clinical guidelines suggest using warfarin for APS-related stroke, but these suggestions are largely based on retrospective studies from the 1990s and expert opinion, rather than high-quality clinical trials. Moreover, the evidence on the role of antiplatelet drugs other than aspirin (e.g., clopidogrel) in APS-related stroke is particularly limited. Considering the relatively young age of patients with APS and the high clinical burden of using warfarin, it is necessary to verify whether warfarin is essential. Thus, the investigators aim to compare clopidogrel-based antiplatelet therapy and warfarin as a secondary preventive medication for patients with APS-related stroke. APS-STROKE is an exploratory, multicenter, prospective, randomized, open, blinded-endpoint clinical trial. Adult patients with definite APS who have a history of ischemic stroke will be included. Patients with high-risk APS (triple positivity or persistently high titers of anti-cardiolipin or anti-β2-glycoprotein I antibodies), systemic lupus erythematous, or indications for continued antiplatelet or anticoagulant therapy will be excluded. Eligible patients will be 1:1 randomized to receive clopidogrel-based antiplatelet therapy or warfarin. Patients assigned to the clopidogrel-based antiplatelet therapy group will be permitted to use additional antiplatelet drugs other than clopidogrel at the investigator's discretion. The primary outcome is a composite of any death, major adverse cardiovascular events, systemic thromboembolic events, and major bleeding during a follow-up period of at least 4 years. This study would provide valuable information for determining the optimal secondary prevention strategy for APS-related stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* History of ischemic stroke (cerebral infarction, transient ischemic attack, or retinal arterial ischemic event)
* Patients who meet the laboratory diagnostic criteria for antiphospholipid syndrome (APS)
* Patients or guardians who agree to the study protocol and sign with informed consent

Exclusion Criteria:

* Patients with high-risk antiphospholipid antibody profile (triple positivity; persistent high-titers exceeding 80 U/mL of anti-cardiolipin or anti-β2 glycoprotein I antibodies)
* Systemic lupus erythematous
* Patients unable to discontinue previously taken anticoagulants or antiplatelet agents (e.g., atrial fibrillation, valvular heart disease, or a history of percutaneous coronary intervention)
* Women who are pregnant, breastfeeding, or intending to become pregnant during the study period
* Deemed unsuitable for participation in the study for more than four years, as per the investigators' discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint | 4 years
  Composite endpoint of any death, major adverse cardiovascular events (MACEs), systemic thromboembolic events, and major bleeding. MACE includes any stroke, transient ischemic attack, and acute coronary syndrome (i.e., ST-elevation myocardial infarction, non-ST elevation myocardial infarction, and hospitalization with unstable angina) in this study. Major bleeding refers to bleeding events meeting the criteria for Bleeding Academic Research Consortium (BARC) type 3 or 5.

SECONDARY OUTCOMES:
MACE | 4 years
  MACE includes any stroke, transient ischemic attack, and acute coronary syndrome (i.e., ST-elevation myocardial infarction, non-ST elevation myocardial infarction, and hospitalization with unstable angina) in this study.
Ischemic stroke | 4 years
  Ischemic stroke or transient ischemic attack
Any bleeding | 4 years
  Major or minor bleeding according to definitions from BARC
Major bleeding | 4 years
  BARC bleeding type 3 or 5
Intracranial bleeding | 4 years
  Intracranial bleeding that is objectively confirmed by brain imaging
Clinically relevant non-major bleeding | 4 years
  Any bleeding that does not fit the criteria for major bleeding but does meet at least one of the following criteria:
  1. requiring nonsurgical, medical intervention by a healthcare professional
  2. leading to hospitalization or increased level of care
  3. prompting evaluation.
Any death | 4 years
  Death from any cause
Thrombosis-related death | 4 years
  Death from arterial, venous, or capillary thrombotic events

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hoon Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (32):
- South Korea (32):
  - Hallym University Sacred Heart Hospital, Anyang
  - Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Jeonbuk National University Hospital, Jeonju
  - Chungnam National University Sejong Hospital, Sejong
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Woman University Seoul Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Uijeongbu Eulji Medical Center, Uijeongbu-si
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miyakis S, Lockshin MD, Atsumi T, Branch DW, Brey RL, Cervera R, Derksen RH, DE Groot PG, Koike T, Meroni PL, Reber G, Shoenfeld Y, Tincani A, Vlachoyiannopoulos PG, Krilis SA. International consensus statement on an update of the classification criteria for definite antiphospholipid syndrome (APS). J Thromb Haemost. 2006 Feb;4(2):295-306. doi: 10.1111/j.1538-7836.2006.01753.x. PMID 16420554
- [Background] Bertero MT, Bazzan M, Carignola R, Montaruli B, Silvestro E, Sciascia S, Vaccarino A, Baldovino S, Roccatello D; Antiphospholipid Piedmont Consortium. Antiphospholipid syndrome in northwest Italy (APS Piedmont Cohort): demographic features, risk factors, clinical and laboratory profile. Lupus. 2012 Jun;21(7):806-9. doi: 10.1177/0961203312446974. PMID 22635240
- [Background] Yang W, Kang MK, Ha SY, Kang DW, Bae J, Lee EJ, Jeong HY, Kim JM, Jung KH, Lee SH. Current status and role of antiphospholipid antibody testing in cryptogenic stroke. Eur J Neurol. 2022 Mar;29(3):753-760. doi: 10.1111/ene.15191. Epub 2021 Dec 3. PMID 34800314
- [Background] Cohen H, Cuadrado MJ, Erkan D, Duarte-Garcia A, Isenberg DA, Knight JS, Ortel TL, Rahman A, Salmon JE, Tektonidou MG, Williams DJ, Willis R, Woller SC, Andrade D. 16th International Congress on Antiphospholipid Antibodies Task Force Report on Antiphospholipid Syndrome Treatment Trends. Lupus. 2020 Oct;29(12):1571-1593. doi: 10.1177/0961203320950461. PMID 33100166
- [Background] Tektonidou MG, Andreoli L, Limper M, Amoura Z, Cervera R, Costedoat-Chalumeau N, Cuadrado MJ, Dorner T, Ferrer-Oliveras R, Hambly K, Khamashta MA, King J, Marchiori F, Meroni PL, Mosca M, Pengo V, Raio L, Ruiz-Irastorza G, Shoenfeld Y, Stojanovich L, Svenungsson E, Wahl D, Tincani A, Ward MM. EULAR recommendations for the management of antiphospholipid syndrome in adults. Ann Rheum Dis. 2019 Oct;78(10):1296-1304. doi: 10.1136/annrheumdis-2019-215213. Epub 2019 May 15. PMID 31092409
- [Background] Keeling D, Mackie I, Moore GW, Greer IA, Greaves M; British Committee for Standards in Haematology. Guidelines on the investigation and management of antiphospholipid syndrome. Br J Haematol. 2012 Apr;157(1):47-58. doi: 10.1111/j.1365-2141.2012.09037.x. Epub 2012 Feb 8. No abstract available. PMID 22313321
- [Background] Rosove MH, Brewer PM. Antiphospholipid thrombosis: clinical course after the first thrombotic event in 70 patients. Ann Intern Med. 1992 Aug 15;117(4):303-8. doi: 10.7326/0003-4819-117-4-303. PMID 1637025
- [Background] Khamashta MA, Cuadrado MJ, Mujic F, Taub NA, Hunt BJ, Hughes GR. The management of thrombosis in the antiphospholipid-antibody syndrome. N Engl J Med. 1995 Apr 13;332(15):993-7. doi: 10.1056/NEJM199504133321504. PMID 7885428
- [Background] Krnic-Barrie S, O'Connor CR, Looney SW, Pierangeli SS, Harris EN. A retrospective review of 61 patients with antiphospholipid syndrome. Analysis of factors influencing recurrent thrombosis. Arch Intern Med. 1997 Oct 13;157(18):2101-8. PMID 9382667
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Pengo V, Denas G, Zoppellaro G, Jose SP, Hoxha A, Ruffatti A, Andreoli L, Tincani A, Cenci C, Prisco D, Fierro T, Gresele P, Cafolla A, De Micheli V, Ghirarduzzi A, Tosetto A, Falanga A, Martinelli I, Testa S, Barcellona D, Gerosa M, Banzato A. Rivaroxaban vs warfarin in high-risk patients with antiphospholipid syndrome. Blood. 2018 Sep 27;132(13):1365-1371. doi: 10.1182/blood-2018-04-848333. Epub 2018 Jul 12. PMID 30002145
- [Background] Erkan D, Barbhaiya M, George D, Sammaritano L, Lockshin M. Moderate versus high-titer persistently anticardiolipin antibody positive patients: are they clinically different and does high-titer anti-beta 2-glycoprotein-I antibody positivity offer additional predictive information? Lupus. 2010 Apr;19(5):613-9. doi: 10.1177/0961203309355300. Epub 2009 Nov 24. PMID 19934177
- [Background] Udry S, Latino JO, Belizna C, Peres Wingeyer S, Fernandez Romero DS, de Larranaga G. A high-risk laboratory profile of antiphospholipid antibodies and thrombosis is associated with a large number of extra-criteria manifestations in obstetric antiphospholipid syndrome. Immunol Res. 2019 Dec;67(6):478-485. doi: 10.1007/s12026-019-09110-x. PMID 31873844
- [Background] Ordi-Ros J, Saez-Comet L, Perez-Conesa M, Vidal X, Riera-Mestre A, Castro-Salomo A, Cuquet-Pedragosa J, Ortiz-Santamaria V, Mauri-Plana M, Sole C, Cortes-Hernandez J. Rivaroxaban Versus Vitamin K Antagonist in Antiphospholipid Syndrome: A Randomized Noninferiority Trial. Ann Intern Med. 2019 Nov 19;171(10):685-694. doi: 10.7326/M19-0291. Epub 2019 Oct 15. PMID 31610549
- [Background] Woller SC, Stevens SM, Kaplan D, Wang TF, Branch DW, Groat D, Wilson EL, Armbruster B, Aston VT, Lloyd JF, Rondina MT, Elliott CG. Apixaban compared with warfarin to prevent thrombosis in thrombotic antiphospholipid syndrome: a randomized trial. Blood Adv. 2022 Mar 22;6(6):1661-1670. doi: 10.1182/bloodadvances.2021005808. PMID 34662890
- [Background] Yang W, Kang DW, Kim JM, Jung KH, Lee SH. Neuroimaging features of antiphospholipid antibody-related stroke compared with atrial fibrillation-related stroke. Sci Rep. 2022 Jul 8;12(1):11686. doi: 10.1038/s41598-022-16019-3. PMID 35804027
- [Background] Kaatz S, Ahmad D, Spyropoulos AC, Schulman S; Subcommittee on Control of Anticoagulation. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26. doi: 10.1111/jth.13140. No abstract available. PMID 26764429
- [Derived] Yang W, Park HK, Koh SH, Kim S, Kim Y, Jung KH, Kang HG, Choi JC, Kim HY, Nam HS, Jeong HS, Kim JT, Kim YS, Yu S, Cho KH, Song TJ, Heo SH, Cho HJ, Sohn SI, Chang Y, Park JM, Oh MS, Kim EG, Shin DI, Kim C, Lee J, Ahn SH, Lee YB, Shin JW, Kim BJ, Kim BJ, Park KY, Kwon HM, Jang H, Kim JM, Kim J, Lee SH; APS-STROKE investigators. Comparison of clopidogrel-based antiplatelet therapy versus warfarin as a secondary prevention strategy for AntiPhospholipid Syndrome-related STROKE (APS-STROKE): Rationale and design of a prospective, randomized, open-label, blinded-endpoint trial. Contemp Clin Trials. 2026 Jan;160:108164. doi: 10.1016/j.cct.2025.108164. Epub 2025 Nov 25. PMID 41308951